CLINICAL TRIAL: NCT07218874
Title: Feasibility and Acceptability of the Remote Oncology Symptom Assessment Application
Acronym: ROSA App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carissa Low, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25070088; R37CA242545 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Solid Tumor Cancer; Chemotherapy
Keywords: quality of life; symptom management; smartphone application
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptom monitoring via smartphone app (Experimental): Participants will rate symptoms daily for 90 days using PRO-CATCAE questions to assess 8 common chemotherapy-related symptoms. Participants will wear a Fitbit (Inspire 3 or similar) for the duration of the study and install the Fitbit app on their smartphone. The Fitbit is a wristwatch-sized waterproof device that assesses heart and breathing rates, physical activity, and sleep, skin temperature, and oxygen levels and wirelessly transmits data to the server.
  Interventions: Behavioral: Mobile Symptom Monitoring and Alert App

INTERVENTIONS:
Behavioral: Mobile Symptom Monitoring and Alert App — Responses range from 0-4; any grade 1 response (reflecting mild symptoms) will trigger a recommendation to view symptom management/education tips available in a self-care library in the app, and any grade 2-4 response (reflecting moderate to severe symptoms) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning symptom. Fitbit data points outside of prespecified thresholds based on physiological norms (for skin temperature and pulse oxygenation) or each participants' historic average (heart rate and activity) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning data point. Reports will be generated and emailed to participants each week displaying summaries/graphs of recent alerts triggered, symptom ratings, and Fitbit data.

SUMMARY:
The goal of this study is to determine whether a mobile application that combines real-time sensor data and patient-reported symptoms to trigger care-team contact recommendations is feasible and beneficial for patients receiving chemotherapy. The main questions it aims to answer are:

* Is the mobile application feasible and acceptable to patients?
* Do the alerts and guidance improve symptom management, quality of life, and engagement with the care team during treatment?

Participants will:

* Complete a demographic questionnaire at the beginning of the study and quality-of-life and health questionnaires at the beginning, midpoint, and end of study.
* Complete daily symptom ratings.
* Wear a Fitbit activity tracker for 90 days.
* At the end of the study, complete a semi-structured interview to provide feedback on the study.
* Optional: At the beginning and end of the study, complete an in-person physical function assessment measuring balance (Short Physical Performance Battery).

DETAILED DESCRIPTION:
Participants (n=50) will be recruited from UPMC Hillman clinics.

If eligible patients consent to participate, they will complete online baseline, midpoint, and end of study questionnaires. Participant's medical records will be reviewed to extract demographic information and clinical covariates, including information about their cancer, its treatment, biological variables such as sex and age, clinical variables such as comorbidities, surgeries and hospitalizations, medications, and other markers of health care utilization (e.g., emergency department visits). Once extracted, these values will be linked only to their study ID number.

Following informed consent, participants will have the ROSA Android or iOS application installed on their smartphones that are capable of running the app (or will be talked through the installation of the app on their smartphone if conducting visit remotely). The application will securely store this information on the device and transmit this information to a secure cloud-based research server over secure network (WiFi or cellular) connection at least once per day. All data will be de-identified and will use only a study ID number linked to identifying participant information in a password protected file. The data captured for the research will not include any personally identifiable information. The data plan requirements of the application are not significantly different from what most smartphone users would require if they use their device to access the Internet for web searching.

At the initial visit (either in person or online, 20-30 minutes), participants will also be oriented to the ecological momentary assessment procedures to assess patient-reported symptoms. Participants will install the ROSA Android or iOS application on their smartphones. The unique non-identifying participant ID will be entered into the app upon initial log in and will be saved locally on the device. This code number will be attached to participant data so that the research team will be able to know which participant code number each survey response is associated with. Participants will be able to set the time of day for which they wish to receive notifications to complete the daily symptom ratings. When participants receive the survey notification, it will open up the study application and they can proceed to take the daily survey (approximately 5 minutes) via an anonymous Qualtrics survey link embedded in the app and opened in their smartphone's internet browser. Symptoms will be assessed using the PRO version of the Common Terminology for Adverse Events (PRO-CTCAE).

Participants will be asked to complete at least one rating per day and will report on symptoms over the last 24 hours. Responses range from 0-4; any grade 1 response (reflecting mild symptoms) will trigger a recommendation to view symptom management/education tips available in a self-care library in the app, and any grade 2-4 response (reflecting moderate to severe symptoms) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning symptom. Reports will be automatically generated and emailed each week displaying their summarized data and a list of all the individual data points that triggered alerts which they can then share with their care team, family members, etc. Weekly reports will include a link to an optional survey asking for feedback on how they've used the last week's report. In addition to the PRO-CTCAE questions in the daily survey, participants will also be asked to rate their overall quality of life for that day from 0 (worst possible) to 10 (best possible), about any cancer treatment they've received since the last survey, about any communication with their cancer care team since their last survey, and approximately how much time they spent each day on tasks related to cancer care.

As feasible, participants will complete the Short Physical Performance Battery (SPPB) at the UPMC Hillman Cancer Center or the research team's office at baseline and at the end of the study. During these visits, this in-person assessment will be administered by trained study team members. Participants that enroll in the study remotely will be invited to complete the in-person SPPB as feasible. The SPPB will be conducted within 2 weeks of the enrollment date and within 2 weeks of the end of study date.

Participants will also be asked to wear a Fitbit device as feasible (Fitbit Inspire 3 or similar) for the duration of the study and to install the Fitbit app on their smartphone. The Fitbit is a wristwatch-sized waterproof device that assesses heart and breathing rates, physical activity, and sleep, skin temperature, and oxygen levels and wirelessly transmits data to the server. Participants will be asked to charge the device as needed, approximately every 7-10 days. If they already own a Fitbit device that collects comparable data to the study provided device, we will request access to their Fitbit data for the duration of their study participation. Fitbit data points outside of prespecified thresholds based on physiological norms (for skin temperature and pulse oxygenation) or each participants' historic average (heart rate and activity) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning data point.

At the end of the study, we will assist participants in removing the ROSA app from their phones. Participants will also complete an end of study interview at this time.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemotherapy at the UPMC Hillman Cancer Center for any solid tumor cancer at any stage with at least two cycles remaining;
* age 18 years or older;
* ability to read and write in English;
* sufficient performance status to participate in research (e.g., Karnofsky performance status of 60-100%); and
* owns and uses an Android smartphone or an iPhone capable of running the study apps.

Exclusion Criteria:

* under 18 years old; and
* unable to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability via semi-structured interviews | At the end of the intervention (at approximately 90 days)
  Post-intervention semi-structured interviews will be conducted to gather participant feedback and assess acceptability of the program (e.g., likelihood to keep using app and to recommend app)
Acceptability via System Usability Scale | At the end of the intervention (at approximately 90 days)
  System Usability Scale (SUS). For odd items, subtract one from the user response. For even-numbered items, subtract the user responses from 5. This scales all values from 0 to 4 (with four being the most positive response). Add up the converted responses for each user and multiply that total by 2.5. Possible range of scores is 0 to 100 representing a composite measure of the overall usability of the system being studied.
Feasibility via accrual rate | From enrollment to the end of the intervention (at approximately 90 days)
  accrual rate (number of participants that enroll [consent and provide at least one form of data] out of number of participants approached)
Feasibility via engagement | From enrollment to the end of the intervention (at approximately 90 days)
  engagement (how many days within the study the participants engaged with the app and had Fitbit data)
Feasibility via completion rate | From enrollment to the end of the intervention (at approximately 90 days)
  completion rate (number of participants that complete the study)

SECONDARY OUTCOMES:
Patient-Reported Physical Symptoms | Change from baseline to the end of the intervention (at approximately 90 days)
  Symptoms will be assessed using the PRO version of the Common Terminology for Adverse Events (PRO-CTCAE; Dueck et al., 2015). PRO-CTCAE questions will assess eight symptoms common during chemotherapy for cancer, including decreased appetite, diarrhea, fatigue, nausea, neuropathy, pain, shortness of breath, and vomiting. The daily PRO-CTCAE questions include conditional branching where participants will not be asked about the severity, frequency, and/or the extent to which a symptom interfered with their activities if they do not endorse that symptom. Participants will be asked to complete at least one rating per day and will report on symptoms over the last 24 hours. Responses range from 0-4, with higher scores indicating more severe symptoms.

OTHER OUTCOMES:
Quality of Life | Change from baseline to the end of the intervention (at approximately 90 days)
  Patient-Reported Outcome Measurement Information System (PROMIS) 29+2 is used to evaluate general health-related quality of life. The seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) have four items per domain and use a 5-point Likert response scale. Possible range of scores for these 7 domains is 4 to 20. The pain intensity item uses a numeric rating scale (0 [no pain] to 10 [worst pain imaginable]). The sum of raw scores for each domain is converted into a standardized T-score using a publicly available conversion table or an online scoring service. Higher scores represent worse symptoms for symptom-oriented domains (anxiety, depression, fatigue, pain intensity, pain interference, and sleep disturbance) and better health outcomes for function-oriented domains (physical functioning and ability to participate in social roles and activities).
Depressive symptoms | Change from baseline to the end of the intervention (at approximately 90 days)
  Center for Epidemiologic Studies Depression Scale (CES-D Scale). Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
Objective physical activity | Change from baseline to the end of the intervention (at approximately 90 days)
  A Bluetooth enabled activity monitor worn throughout the study will estimate number of steps/day.
Activity disruption | Change from baseline to the end of the intervention (at approximately 90 days)
  Sickness Impact Profile short form (6 items) is used to assess a person's perception of their health status with respect to their disease impact. Possible range of scores is 0 (0%) to 6 (100%). Higher scores represent poor health status or a major impact of illness on behavior.
Instrumental Support | Change from baseline to the end of the intervention (at approximately 90 days)
  PROMIS Instrumental Support v2.0 - Short Form 4a is 4-item short form assessing perceived availability of assistance with material, cognitive or task performance. Responses are rated on a 5-point Likert scale, yielding a total score range of 4 to 16. Higher scores indicate greater perceived instrumental support.
Self-Efficacy for Managing Symptoms | Change from baseline to the end of the intervention (at approximately 90 days)
  PROMIS Self-Efficacy for Managing Symptoms v1.0 - Short Form 4a is a 4-item short form assessing confidence to manage/control symptoms, to manage symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships, or recreational activities. Responses are rated on a 5-point Likert scale, yielding a total score range of 4 to 16. Higher scores indicate greater perceived self-efficacy for managing symptoms.
Short Physical Performance Battery (SPPB) | Change from baseline to the end of the intervention (at approximately 90 days)
  The SPPB is a short battery of performance tests of lower extremity functioning. The tests measure gait speed, standing balance, and lower extremity strength and power. To test gait speed, patients are instructed to walk an 8-foot walking course at their usual pace with assistive devices if needed. Four progressively more challenging positions are used to test balance (bipedal [feet next to each other], semi-tandem [one foot slightly in front of the other], and full tandem [one foot in front of the other]). To test lower extremity strength, patients are asked to stand up and sit down five times as quickly as possible and are timed from the initial sitting position to the final standing position at the end of the fifth stand. Each component (gait speed, balance, chair stands) is scored 0-4, where 0 is unable to complete task and 4 indicates highest level of performance. Total score is 0-12 with higher scores indicating better lower extremity function.
Patient-Centered Communication Questionnaire - Cancer | Change from baseline to the end of the intervention (at approximately 90 days)
  The PCC-Ca-36 is a 36-item questionnaire to assess patients' experience with patient-centered communication during cancer care. It evaluates 6 core functions: exchanging information, fostering healing relationships, making decisions, attention to emotions, taking care of yourself, and dealing with uncertainty. Responses are rated on a 5-point Likert scale with some items having the option "Does not apply". Individual functions are scored by averaging items within the function and an overall PCC score is the average of all items. Higher scores indicate better perceived patient-centered communication.

CONTACTS AND LOCATIONS:
Overall Officials: Carissa A Low, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Preliminary IPD data from this pilot study will not be shared